CLINICAL TRIAL: NCT06681558
Title: Comparison of Procedural Oxygen Mask vs. Conventional Nasal Cannula for Hypoxemia Prevention During Endoscopic Retrograde Cholangiopancreatography (ERCP): A Randomized Controlled Trial
Brief Title: Procedural Oxygen Mask vs. Nasal Cannula for Hypoxemia Prevention During Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Bedirhan Günel, Principal Investigator, Kocaeli City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KSH-ANREA-BG-03
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Hypoxemia
Keywords: Hypoxemia; Endoscopic Retrograde Cholangiopancreatography; Airway Management; Sedation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group Nasal Cannula (Active Comparator): Oxygen will be administered to this group via a conventional nasal cannula.
  Interventions: Device: Group Nasal Cannula
- Group Procedural Oxygen Mask (Active Comparator): Oxygen will be administered to this group via a Procedural Oxygen Mask.
  Interventions: Device: Group Procedural Oxygen Mask

INTERVENTIONS:
Device: Group Nasal Cannula — Oxygen administered during the endoscopic retrograde cholangiopancreatography (ERCP) procedure will be delivered through a conventional oxygen mask.
  The nasal cannula is a device that provides oxygen to patients through the nasal passages.
  Arms: Group Nasal Cannula
Device: Group Procedural Oxygen Mask — Oxygen administered during the endoscopic retrograde cholangiopancreatography (ERCP) procedure will be delivered through a Procedural Oxygen Mask (POM® ELITE MF). The procedural oxygen mask is a device that covers both the mouth and nose to deliver oxygen to the patient. Its reservoir feature increases the concentration of delivered oxygen
  Arms: Group Procedural Oxygen Mask

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an imaging procedure that visualizes the drainage ducts of the pancreas, gallbladder, and liver through the use of a duodenoscope and contrast media. By endoscopically identifying the ampulla of Vater, the common bile duct is cannulated. ERCP is also frequently utilized for therapeutic interventions, such as endoscopic sphincterotomy, bile duct stone extraction, stent placement in malignant and benign biliary strictures, and biopsy collection, thus playing a critical role in both the diagnosis and treatment of pancreatobiliary disorders.

ERCP, being more invasive than routine upper endoscopies or colonoscopies, typically necessitates deeper levels of sedation. The procedure is performed in the prone, modified prone, or lateral decubitus position, which increases the risk of hypoxemia and hypoventilation due to upper airway obstruction. Furthermore, endoscopic instruments inserted through the oral cavity limit anesthesiologists' access to the patient's airway, thereby restricting ventilation support during gastrointestinal endoscopy. Ensuring airway stability during sedation is paramount for patient safety and procedural efficacy. Currently, a range of devices, including traditional nasal cannulas, high-flow oxygen masks, and procedural oxygen masks, are routinely employed to provide oxygen support throughout the procedure.

The existing literature includes randomized controlled trials and systematic reviews aimed at preventing hypoxemia during ERCP. Through this study, investigators aim to make a novel contribution to the literature by assessing the effectiveness of a recently introduced procedural oxygen mask.

DETAILED DESCRIPTION:
This study aims to compare the efficacy of different oxygen delivery methods (Nasal Cannula [NC] and Procedural Oxygen Mask [POM]) in preventing the incidence of hypoxemia during Endoscopic Retrograde Cholangiopancreatography (ERCP). Designed as a randomized controlled prospective study, participants were assigned into two groups, Group N (NC) and Group P (POM), at a 1:1 ratio through randomization. The randomization was performed using computer-assisted random allocation; however, due to the visual differences in the oxygen delivery devices, neither healthcare providers nor patients could be blinded to the randomization results. A power analysis conducted to establish a statistical power of 80% and an alpha level of 0.05 indicated that a total of 140 patients, with 70 patients in each group, should be included in the study. Considering potential dropouts, 150 patients will be included in the study This evaluation ensures that an adequate sample size is obtained to detect a significant difference in the incidence of hypoxemia.

Throughout the ERCP procedure, all patients will be monitored using pulse oximetry, electrocardiography (ECG), and non-invasive blood pressure monitoring. Capnography will be applied in both groups, and necessary interventions will be carried out by anesthesia specialists if a patient's oxygen saturation falls below 90%. All interventions and events will be meticulously documented. Following the procedure, patients will be monitored in the post-anesthesia care unit (PACU), and those with a Post-Anesthesia Discharge Scoring System (PADSS) score of 9 or higher will be discharged.

Anesthesia Management The oxygen flow rate will be maintained constant throughout the procedure. Initially, patients will receive midazolam at a dose of 0.02 mg/kg, followed by 0.3 mg/kg of ketamine. To ensure sedation, propofol will be administered as an initial bolus dose of 0.5-1.0 mg/kg; further bolus doses of 0.25-0.5 mg/kg will be given every 1-3 minutes to maintain the desired sedation level. The target sedation level will be aimed at 3-4 on the Ramsay Sedation Scale (RSS), and these target values will be preserved during the procedure. Upon completion of the procedure, patients will be awakened using verbal and tactile stimuli; once the RSS reaches 2, they will be transferred to the PACU. In the PACU, patients will be discharged if they achieve a PADSS score of 9 or above.

Oxygen Reserve Index (ORi) measurement will performed on all patients. The ORi value will measured and recorded at the plateau level during the preoxygenation stage (as the baseline), immediately after the start of the procedure, at the end of the procedure, and the highest ORi value measured throughout the procedure

Vital signs, procedure durations, and dosages of medications used for each patient will be meticulously recorded. All anesthesia-related decisions during the procedure will be made by the supervising anesthesia specialist.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* American Society of Anesthesiologists (ASA) classification of 1-2-3
* Patients scheduled for ERCP at Kocaeli City Hospital Endoscopy Unit

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients with allergies to ketamine, propofol, or midazolam
* Patients diagnosed with psychiatric disorders
* Patients with a body mass index (BMI) >30 kg/m²
* Patients with cognitive impairment, dementia, or communication issues
* Pregnant patients or those in the postpartum period
* Patients diagnosed with sleep apnea syndrome
* History of intubation within the last 3 months
* History of lower respiratory tract infection within the last 3 months
* History of intensive care unit admission within the last 3 months
* Patients with a tracheostomy
* Patients with a history of tracheostomy
* Patients who are oxygen-dependent due to a medical condition
* Patients with lung cancer or who have undergone surgery on their lungs
* Patients with asthma, COPD, or interstitial lung diseases
* Patients with uncontrolled hypertension (BP >180/110)
* Patients receiving home care

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
incidence of hypoxemia | Continuous SpO2 monitoring will be performed throughout the ERCP procedure
  The incidence of hypoxemia during sedation (defined as SpO2 < 90%). SpO₂ will be continuously measured using a pulse oximeter (GE Healthcare) to monitor and record oxygen saturation levels throughout sedation.

SECONDARY OUTCOMES:
Number of hypoxemia episodes | Continuous SpO2 monitoring will be performed throughout the ERCP procedure
  An episode was recorded when SpO2 dropped below 90% after reaching a level of SpO2 ≥ 90% for 30 seconds. SpO₂ will be continuously measured using a pulse oximeter (GE Healthcare) to monitor and record oxygen saturation levels throughout sedation.
Duration of hypoxemia | Continuous SpO2 monitoring will be performed throughout the ERCP procedure
  Defined as the time taken to reach SpO2 ≥ 90%. SpO₂ will be continuously measured using a pulse oximeter (GE Healthcare) to monitor and record oxygen saturation levels throughout sedation.
Minimum SpO2 value observed during the procedure | Continuous SpO2 monitoring will be performed throughout the ERCP procedure
  Minimum SpO2 value observed during the procedure. SpO₂ will be continuously measured using a pulse oximeter (GE Healthcare) to monitor and record oxygen saturation levels throughout sedation.
Oxygen Reserve Index (as the baseline) | Continuous Oxygen Reserve Index monitoring will be performed after prepreoxygenation
  The Oxygen Reserve Index (ORi) value will be measured at the plateau level during the preoxygenation stage (as the baseline)
Oxygen Reserve Index (immediately after the start of the procedure) | Continuous Oxygen Reserve Index monitoring will be performed throughout the ERCP procedure
  Oxygen Reserve Index (immediately after the start of the procedure) value will bemeasured
Oxygen Reserve Index (at the end of the procedure) | Continuous Oxygen Reserve Index monitoring will be performed throughout the ERCP procedure
  Oxygen Reserve Index (at the end of the procedure) value will be measured
Oxygen Reserve Index (highest ORi value will be measured) | Continuous Oxygen Reserve Index monitoring will be performed throughout the ERCP procedure
  Oxygen Reserve Index (highest ORi value will be measured) value will be measured
airway management | Interventions related to airway management causing interruptions during the procedure
  This measure will assess the frequency and types of airway management interventions performed during the procedure that result in interruptions. The specific interventions include chin lift, jaw thrust, mask ventilation, need for aspiration, and repositioning of the nasal cannula or Procedural Oxygen Mask (POM). Data will be collected through direct observation and recorded in the procedural notes, capturing the number of times each intervention was required.
Other potential complications | during the procedure
  Other potential complications that may arise during the procedure (hypotension, hypertension, bradycardia, tachycardia, movements that hinder the procedure) (Hypotension is defined as a decrease in the patient's baseline systolic blood pressure of more than 20% or a drop below 90 mm Hg. Hypertension is defined as an increase in the patient's baseline systolic blood pressure of more than 20%. A heart rate below 60 beats per minute is considered bradycardia, while a rate above 100 beats per minute is classified as tachycardia).
Number of Participants with Early Termination of Procedure Due to Sedation | during the procedure
  This measure will track the number of participants for whom the procedure was terminated early as a result of sedation-related factors.
ERCP duration | up to 60 minutes (or the estimated average duration of the procedure)
  defined as the time from the start of the procedure until the gastroscope is completely removed.
Recovery time | up to a maximum of 90 minutes (or the estimated average recovery time for the procedure)
  defined as the time from the administration of the first anesthetic until the procedure is completely finished and Ramsey Sedation Scale (RSS) reaches 2.
Discharge time | assessed during the recovery period, up to a maximum of 120 minutes (or the estimated average time for the procedure recovery)
  defined as the time from the removal of the gastroscope until MPADS is 9 or above
Gastroenterologist satisfaction | with data reported immediately following the completion of the procedure.
  a 10-point scoring system was used, where 0 indicates "unmanageable, numerous interruptions or terminated procedure," and 10 indicates "excellent sedation, no interruptions"
Postoperative nausea, vomiting, pain, aspiration, and other potential complications | Data will be recorded until discharge from the PACU, which is expected to occur within up to 2 hours after the procedure."
  Postoperative nausea, vomiting, pain, aspiration, and other potential complications
Patient satisfaction related to anesthesia | Data will be recorded until discharge from the PACU, which is expected to occur within up to 2 hours after the procedure."
  Patient satisfaction related to anesthesia was assessed and recorded before discharge (a scale from 0 to 10 was used, where 0 means "very poor, I would never undergo this procedure again," and 10 means "excellent, I would undergo this procedure again in the same manner").

CONTACTS AND LOCATIONS:
Overall Officials: BEDİRHAN GÜNEL, MD, Study Chair — Kocaeli City Hospital; AYŞE ŞENCAN, MD, Principal Investigator — Kocaeli City Hospital; YASEMİN Y. TAVŞANOĞLU, MD, Principal Investigator — Kocaeli City Hospital; ZEKİ İSLAMOĞLU, MD, Principal Investigator — Kocaeli City Hospital; AHMET YÜKSEK, ASSOC. PROF, Principal Investigator — Kocaeli City Hospital; MEHMET YILMAZ, ASSOC.PROF, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, İ̇zmi̇t, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal data and study data will not be shared.

REFERENCES:
- [Derived] Gunel B, Sencan A, Tavsanoglu ZY, Cevik T, Atli E, Islamoglu Z, Yuksek A, Yilmaz M. Comparison of Procedural Oxygen Mask Versus Conventional Nasal Cannula for Hypoxemia Prevention During Endoscopic Retrograde Cholangiopancreatography: A Randomized Controlled Trial. Dig Dis Sci. 2025 Dec;70(12):4281-4291. doi: 10.1007/s10620-025-09264-9. Epub 2025 Jul 30. PMID 40736944